CLINICAL TRIAL: NCT06032650
Title: Calisthenics Versus High-intensity Interval Exercises on Health-related Outcomes in Patients With Non-alcoholic Fatty Liver
Brief Title: Calisthenics Versus High Intensity Interval Training in NAFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Younis Mahmoud Abdel-Salam, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004531
Record Dates: First submitted 2023-09-03; First posted 2023-09-13 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD , Calisthenics , High intensity interval training
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group A (Calisthenics exercise) (Experimental): Group (A) (n =30) will receive calisthenics exercise three times /week for eight weeks, patients in this group will receive four forms of calisthenics exercise (squats, curl up, push up, blank) starting free and upgrading intensity according to ability of the patients.
  Interventions: Other: Calisthenics exercise and High intensity interval training
- Study group B (High intensity interval training) (Experimental): Group (B) (n =30) will receive high intensity interval training three times /week for eight weeks, A motorized treadmill device (KETTLER, laufband alpha run 600, German) with a minimum speed of 0.5km/hr and capability to display the distance in kilometer per hour will be used in this study. Intensity of HIIT will be measured using Bruce protocol to calculate target heart rate of each patient.
  Interventions: Other: Calisthenics exercise and High intensity interval training

INTERVENTIONS:
Other: Calisthenics exercise and High intensity interval training — 1. The calisthenics exercise focuses on big muscles and can be combined with breathing exercises and applied rhythmically,10-15 for each exercise,1-3 sets,3 days/week for 8 weeks. It will be progressed gradually by increasing the number of sets, repetitions and by using elastic bands and weighted vest progression.
  2. High intensity interval training will be on treadmill for eight weeks, three times/week based on the following program:-Warming up period for 5 min at intensity corresponding to 65-75% of heart rate maximum (HRmax).Training phase for 30 min divided into four sets of 4-min length each at intensity equals 85- 90% of HRmax interspersed by 3 minutes low intensity walking at the level of 65-75% of HRmax.Cooling down period for 5 min of at 50-60% of the HRmax

SUMMARY:
According to sample size calculation and after achieving the inclusion criteria, sixty patients with non-alcoholic fatty liver (NAFL) of both genders will be enrolled in this study and their ages will be ranged from30s-40s; they will be selected from internal medicine-outpatient clinics, Cairo University Hospitals; they will participate in the study for 8 weeks, and randomly be assigned into two equal groups in number.

Group (A) (n =30) will receive calisthenics exercise three times /week for eight weeks, group (B) (n =30) will receive HIIT for three times /week for eight weeks and all patients in both groups will receive their prescribed medication (Statin 5mg ).

DETAILED DESCRIPTION:
A) Evaluation equipment:

All patients will be evaluated before and after treatment protocol.

1. Body composition analyzer (in body 230):- It will be used for estimating body composition, to measure the percentage of the body free fat mass, lean body mass and body mass index (BMI).

   Fig (1) Body composition analyzer (in body 230)
2. Mercury and digital sphygmomanometer and stethoscope: it will be used to measure blood pressure. (Niscomed PW-216)
3. Pulse oximeter: It will be used to monitor heart rate and oxygen saturation continuously during exercise (SantaMedical Generation 2 Fingertip).

   Fig (2) Pulse oximeter
4. Bruce protocol:-to assess functional capacity (Vo2) max and intensity of exercise.
5. Tape measurement: - to assess waist circumference, waist / hip ratio.
6. Clini-chem 2 analyzer: - to analyze blood lipid profile and liver enzymes.

   Fig (3) Clini-chem 2 analyzer
7. Abdominal Ultrasonography (USG) (Siemens, ACUSON NX3 ELITE, and German):- to measure size of the liver, thickness of fat outside liver, as well as severity of the fat infiltration.
8. International Physical Activity Questionnaire-Short Version (IPAQ)):- to assess level of physical activity that patients do as part of their daily lives.
9. Borg scale: - to estimate effort, exertion, breathlessness and fatigue during physical work.

B. Training equipment:-

* A motorized treadmill device (KETTLER, laufband alpha run 600, German) with a minimum speed of 0.5km/hr and capability to display the distance in kilometer per hour will be used in this study.
* Weighted vest progressions and elastic bands: - for calisthenics exercise. -Procedure of the study:- -Assessment procedure:-

A) History and physical examination:

Complete history taking will be conducted to collect data about patient's general condition, physical activity, current medication, and measuring blood pressure.

B) Anthropometric measurement:

1. Body composition analysis: - By using body composition analyzer device (In body 230). The patient will put off his shoes and socks and stand on the device. The device measures his weight and height automatically then the patient will hold the arms of the device to measure total body fat (free fat mass), lean mass and body mass index (BMI). Free fat mass (FM) % 18-24%for men; 25-31%for women and lean mass (LBM) for men 76-82%; for women 69-75% according to The American Council on Exercise (ACE) .
2. Waist circumference (WC) and Waist to hip ratio (WHR):-: Placing a tape horizontal in the midpoint between iliac crest and last rib, and take the measure just after expiration.

Hip circumference will be measured from the widest point of the hip; then dividing waist circumference by hip circumference to calculate waist to hip ratio. According to world health organization, normal cut off values of waist circumference (WC < 88 cm for men; WC < 102 cm or less for women) and waist to hip ratio (WHR < .95 cm for men ; WHR < .80 cm for women).(World Health Organization .2000) 3- Functional capacity (VO2 max):- Using Bruce protocol for multistage treadmill testing of maximal exercise testing will be used as the following 3-min stages: Stage I (2 mph, 10% grade), Stage II (2.5 mph, 12% grade), Stage III (3.4 mph, 14% grade), and Stage IV (4.2 mph, 16%). (Bruce et al., 1963) VO2 max will be estimated from treadmill time based on following equation: For Men VO2 max = 14.8 - (1.379 x T) +(0.451 x T²) - (0.012 x T³) For Women VO2 max = 4.38 x T - 3.9 T = Total time on the treadmill measured as a fraction of a minute i.e.: A test time of 9 minutes 30 seconds would be written as T=9.5 .(Khurana and Oommen 2016) C) Liver enzymes analysis:- According to American Gastroenterological association ,the normal values of liver enzymes (alanine amino transferase ( ALT) 7-55 U/L, aspartate aminotransferase (AST) 8-48 U/L ,gamma glutamyl transferase (GGT) 9-85U/L ). (American Gastroenterological association. 2002)

D) Blood lipid profile analysis:- According to The National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III), the normal reference range of lipid profile (total cholesterol < 200 mg\dl, low- density lipoprotein cholesterol (LDL-C) <100 mg\dl, triglyceride (TG) <150 mg\dl, high density lipoprotein cholesterol (HDL-C) ≥60mg\dl, LDL/HDL3.5/1 mg\dl). (Cleeman et al., 2001) E) Abdominal Ultrasonography (USG):- A 10 MHZ sonosite 180 plus US sanner (penetration depth of 2.2 cm) will be used, Ultrasonographic findings in the liver will be as the following:-

* Increase in hepatic echogenicity.
* Decreased penetration of the deep part of the liver.
* Decreased echogenicity of the diaphragm and intrahepatic portal vessels. (Ma et al., 2011)

F) The International Physical Activity Questionnaire-Short Version (IPAQ)):-It is self - report questionnaire, It consists of seven Open-ended questions surrounding individuals' last seven-day recall of physical activity. The IPAQ records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. Appendix II G) Borg scale: - It is a scale of 0-10;. The scale will allow individuals to subjectively rate their level of exertion during exercise or exercise testing. Appendix III (2) Treatment procedure:- Group (A):- that included 30 non-alcoholic fatty liver patients will participate in calisthenics exercise for eight weeks, Three times/week based on the following program:-

Exercise prescription:

* Mode of exercise: Strengthening exercise.
* Modality of exercise: Bodyweight exercises and require little equipment.
* Forms of exercises:

  1. Sit-Ups that work on Lower abs, mid abs, upper abs, hip flexors, chest, shoulders, quads, and hamstrings.

     Fig (4) Sit -up exercise
  2. Push-Ups that work on Pectorals (chest), biceps, lats, back and core.

Fig (5) Push-up exercise

3- Plank:-That works on abs, shoulders, back, core and glutes,

Fig (6) Plank exercise

4- Squats that work on quads, hamstring, glutes, lower abs and core.

Fig (7) squat exercise

* Repetitions: 10-15 for each exercise.
* Sets: 1-3 sets.
* Intensity of exercise: Moderate-intensity strength exercise training (65%-85%) of (HRmax). (Guzel et al .,2012 )
* Duration: 5-10 minutes warming-up in the form of simple stretching exercises .This is followed by the active phase (20 to 30 minutes) during which a 5-10 seconds passive rest will be allowed in-between repetitions and 1-2 minute passive recovery will be permitted in-between sets. There will be also a cooling down phase for 5 minutes simple stretching exercises.
* Frequency: 3 days/week for 8 weeks.
* Progression: the exercise program will be progressed gradually by increasing the number of sets, repetitions and by using elastic bands and weighted vest progression.

Group (B): that included 30 non-alcoholic fatty liver patients will participate in high intensity interval training on treadmill for eight weeks, three times/week based on the following program:-

1. Warming up period for 5 min at intensity corresponding to 65-75% of heart rate maximum (HRmax).
2. Training phase for 30 min divided into four sets of 4-min length each at intensity equals 85- 90% of HRmax interspersed by 3 minutes low intensity walking at the level of 65-75% of HRmax.
3. Cooling down period for 5 min of at 50-60% of the HRmax. (El-Deeb et al., 2018)

All patients will be trained at the lower intensity limit for the first 2 weeks of the program before increasing the intensity levels toward the upper limit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sixty patients with non-alcoholic fatty liver disease (NAFLD) of both genders.

  2. Patients with mild non-alcoholic fatty liver disease (NAFLD) according to ultrasonography fatty liver indicator (US-FLI) score (2-4).( Chen et al.,2020) 3. Their age will be ranged from 30s-40s. 4. Body mass index (BMI) from 30 to 34.9 kg/m2. 5. Body free fat mass (FFM) percentage > 25 % for men,> 35 % for women. 6. Lean body mass (LBM) parentage < 76 % for men; < 69% for women. 7. Waist circumference ≥ 102 cm for men, > 88 cm for women. 8. Waist/Hip ratio > 0.9% for men and > 0.8% for women. 9. Elevated liver enzymes (ALT> 55 U/L, AST> 48 UL, GGT>85 U/L, AST/ALT <1 U/L).

  10. Patient with dyslipidemia who has one or more from the following blood lipid values (total cholesterol > 200 mg\dl, LDL > 130 mg\dl, TG >150 mg\dl, HDL< 40mg\dl or LDL/HDL ratio > 4).

  11. Low levels of physical activity (using the International Physical Activity Questionnaire- Short Version (IPAQ)) ≤ 10 min walking per day.

  12. Liver size estimated by ultrasonography more than 5% from the normal liver size without hepatocellular damage.

Exclusion Criteria:

* The patient will be excluded if he has one of the following:-

  1. Unstable cardiovascular problems like arrhythmia and heart failure.
  2. Active Hepatitis C virus HCV.
  3. Diabetes mellitus (DM).
  4. Hypertensive patients (>140/90mmHg).
  5. Active Smoker.
  6. Chronic chest disease.
  7. Patients on medications affecting muscle power as steroids.
  8. Auditory and visual problems.
  9. Pregnancy & lactation.
  10. Clinically significant peripheral vascular disease (ABPI < 80 %).
  11. Patients who take beta-blockers.
  12. Severe anemia.
  13. Patients with chronic renal failure.
  14. Musculoskeletal or neurological limitation to physical exercise.
  15. Any cognitive impairment that interferes with prescribed exercise procedures.
  16. .Participation in regular exercise training of any type in the previous 3 months

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Liver ultrasound parameters | up to 8 weeks
  Ultrasonography (USG) (Siemens, ACUSON NX3 ELITE, and German):- to measure size of the liver, thickness of fat outside liver, as well as severity of the fat infiltration
  Ultrasound :-(Siemens, ACUSON NX3 ELITE, and German):- to measure size of the liver, thickness of fat outside liver, as well as severity of the fat infiltration
Blood lipid profile | up to 8 weeks
  Cholosterol,TAG,HDL,LDLand LDL/HDL ratio

SECONDARY OUTCOMES:
Body composition analyzer | up to 8 weeks
  In body 230:- It will be used for estimating body composition, to measure the percentage of the body free fat mass, lean body mass and body mass index (BMI).
Waist circumference(WC) and waist hip ratio(WHR) | up to 8 weeks
  Placing a tape horizontal in the midpoint between iliac crest and last rib, and take the measure just after expiration.
  Hip circumference will be measured from the widest point of the hip; then dividing waist circumference by hip circumference to calculate waist to hip ratio. According to world health organization, normal cut off values of waist circumference (WC < 88 cm for men; WC < 102 cm or less for women) and waist to hip ratio (WHR < .95 cm for men ; WHR < .80 cm for women
Functional capacity (VO2)Max | up to 8 weeks
  Using Bruce protocol for multistage treadmill testing of maximal exercise testing will be used as the following 3-min stages: Stage I (2 mph, 10% grade), Stage II (2.5 mph, 12% grade), Stage III (3.4 mph, 14% grade), and Stage IV (4.2 mph, 16%). (Bruce et al., 1963) VO2 max will be estimated from treadmill time based on following equation: For Men VO2 max = 14.8 - (1.379 x T) +(0.451 x T²) - (0.012 x T³) For Women VO2 max = 4.38 x T - 3.9 T = Total time on the treadmill measured as a fraction of a minute i.e.: A test time of 9 minutes 30 seconds would be written as T=9.
Physical activity level | up to 8 weeks
  to assess level of physical activity that patients do as part of their daily lives by using International Physical Activity Questionnaire-Short Version (IPAQ))
Level of exertion and fatigue | up to 8 weeks
  By using borg scale: - to estimate effort, exertion, breathlessness and fatigue during physical work.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Y mahmoud, AI, Principal Investigator — faculty of physical therapy; NESREEN G EL-NAHAS, Professor, Study Chair — faculty of physical therapy; Hend A ABD EL-MONAEM, Lecturer, Study Director — faculty of physical therapy; KHALED Y MOHAMED, Professor, Study Director — National research center; MOHAMED K MITKES, Researcher, Study Director — National research center
Locations (1):
- Fatma Younis Mahmoud, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelbasset WK, Tantawy SA, Kamel DM, Alqahtani BA, Soliman GS. A randomized controlled trial on the effectiveness of 8-week high-intensity interval exercise on intrahepatic triglycerides, visceral lipids, and health-related quality of life in diabetic obese patients with nonalcoholic fatty liver disease. Medicine (Baltimore). 2019 Mar;98(12):e14918. doi: 10.1097/MD.0000000000014918. PMID 30896648
- [Background] BRUCE RA, BLACKMON JR, JONES JW, STRAIT G. EXERCISING TESTING IN ADULT NORMAL SUBJECTS AND CARDIAC PATIENTS. Pediatrics. 1963 Oct;32:SUPPL 742-56. No abstract available. PMID 14070531
- [Background] American Gastroenterological Association. American Gastroenterological Association medical position statement: evaluation of liver chemistry tests. Gastroenterology. 2002 Oct;123(4):1364-6. doi: 10.1053/gast.2002.36060. No abstract available. PMID 12360497
- [Background] Brunner KT, Henneberg CJ, Wilechansky RM, Long MT. Nonalcoholic Fatty Liver Disease and Obesity Treatment. Curr Obes Rep. 2019 Sep;8(3):220-228. doi: 10.1007/s13679-019-00345-1. PMID 30945129
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183